CLINICAL TRIAL: NCT00719134
Title: The Effects of Expectation and Knowledge on Rizatriptan and Placebo Treatment of Acute Migraine Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Rami Burstein, Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2007-P-000220
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Episodic Migraine
MeSH Terms: interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Maxalt administration at onset of migraine
  Interventions: Drug: Maxalt
- 2 (Placebo Comparator)
  Interventions: Drug: placebo pill
- 3 (Experimental)
  Interventions: Drug: Maxalt
- 4 (Placebo Comparator)
  Interventions: Drug: placebo pills
- 5 (Experimental)
  Interventions: Drug: Maxalt
- 6 (Experimental)
  Interventions: Drug: placebo pills

INTERVENTIONS:
Drug: Maxalt — anti-migraine drug
  Other Names: rizatriptan
  Arms: 1; 3; 5
Drug: placebo pill — placebo pills
  Arms: 2
Drug: placebo pills — placebo pills
  Arms: 4; 6

SUMMARY:
Evidence-based medicine depends on distinguishing between pharmacological effects and placebo effects in randomized controlled trials (RCT). This proposal seeks to rigorously investigate fundamental questions concerning pharmacological effects, placebo effects and their interactions. Relief of symptoms of acute migraine will be the test condition for this scientific experiment because of migraine's evident clinical significance and the possibility of using participants as their own control during sequential acute migraine attacks. Our overall goal is to elucidate how the pharmacological effects of 100 mg rizatriptan (an FDA-proven effective medication for acute migraine) and the effects of placebo treatment can be modified by varied knowledge and/or expectation ("contextual") conditions. Such knowledge has the possibility to suggest potentially more efficient methodologies to test new medications that can be used to augment and enhance the apparatus of the RCT.

General Aim: To elucidate and clarify what is a pharmacological effect and what is a placebo effect, how such effects vary in different knowledge/expectations contexts, and mutually constitute one another and interact.

General Hypothesis: The measured pharmacological effect of an effective medication (rizatriptan) and the measured effect of placebo treatment are determined significantly by different knowledge/expectations contexts.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered for this study if they suffer from classical or common migraine for at least 3 years.
* Candidates will recruited from the clinical case load of Dr. Zahid Bajwa and the headache and pain management center at BIDMC.
* Only patients older than 18 years of age,
* Able to communicate clearly in English,
* Able to give an informed consent will be considered as candidates.
* No limitation of gender or race is justified and thus, it is open to all patients fulfilling criteria for migraine type headache.
* Patients will be able to withdraw from the study at any time.
* They will be included in the study if they meet the criteria for migraine with or without aura (Headache-classification-committee-of-the-International-Headache-Society 1988), if they had >4 migraine attacks each month for the previous year.

Exclusion Criteria:

* Exclusion criteria will include cardiovascular or cerebrovascular disorders,
* Cardiac risk factors and liver disease,
* Uncontrolled hypertension,
* Peripheral and central nervous system disorders that affect sensory functions (such as sensory neuropathies and chronic pain),
* The use of opiates or other analgesic drugs for any reason, and the use of other prophylactic anti-migraine drugs.
* Any patient with active hepatitis or elevated liver enzymes (based on their BIDMC medical record) will be excluded as well.
* Employees who are under the direct supervision of the investigators will not participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Burstein, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Pain Clinic at Beth Israel Deaconess Medical Center, Brookline, Massachusetts, United States

REFERENCES:
- [Result] Kam-Hansen S, Jakubowski M, Kelley JM, Kirsch I, Hoaglin DC, Kaptchuk TJ, Burstein R. Altered placebo and drug labeling changes the outcome of episodic migraine attacks. Sci Transl Med. 2014 Jan 8;6(218):218ra5. doi: 10.1126/scitranslmed.3006175. PMID 24401940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 98 persons pre-screened for eligibility between December 2008 and March 2010, 19 were excluded and 3 declined to participate. The remaining 76 persons signed the consent form, but 10 of them dropped out of the study for various reasons. Participants were recruited from Beth Israel Deaconess Medical Center outpatient clinics.
Pre-assignment Details: Reasons for excluding 19 of the pre-screened subjects include chronic migraine, chronic daily headache, tension type headache, fibromyalgia, daily use of opioids, and medication overuse headache. We randomized participants to one of 8 treatment sequences and each patient received 3 treatments with Maxalt and 3 treatments with Placebo.
Groups:
- All Participants: 76 subjects were randomized to 8 different treatment sequences. Each sequience included treating 6 attacks. 66 subjects completed their treatment assignment.
Period: Overall Study
Arm/Group | All Participants
Started | 76
Completed | 66
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 76
Headache intensity [Mean (Standard Deviation); unit: units on a scale] — pain score at 30 minutes after onset of migraine as measured on a visual analog scale that ranges from 0 (no pain) to 10 (worst pain imaginable).
  units on a scale | 4.6 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Headache Intensity
Description: The primary outcome measure was the change in headache between the baseline pain score recorded 30 min after the onset of headache and the pain score recorded 2 hours later as measured on a visual analog scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: 2 hours after treatment
Population: For the primary endpoint, change in headache intensity from baseline to 2 hours after treatment, we used generalized linear mixed models with a normal random component and a logarithmic link function to analyze the pain scores.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | All Participants
Number analyzed (Participants) | 66
percent change
  percent change with Maxalt | -47.6 [-53.0 to -41.5]
  percent change with placebo | -20.7 [-26.7 to -14.3]

2. Secondary Outcome: Pain Free at 2 Hours After Treatment
Description: A secondary measure of attack outcome was based on categorical classification of the pain freedom (pain score = 0) 2.5 hours after onset of headache.
Time Frame: 2 hours after treatment
Population: For the secondary endpoint, the proportion of patients who were free from pain 2 hours after treatment, we used a mixed-effects logistic regression model to analyze the individual dichotomous outcomes.
Measure: Number (95% Confidence Interval); unit: percent of patients pain free
Arm/Group | All Participants
Number analyzed (Participants) | 66
percent of patients pain free
  pain free with maxalt | 25.5 [17.2 to 36.2]
  pain free with placebo | 6.6 [3.4 to 12.2]

ADVERSE EVENTS:
Arm/Group | Maxalt | Placebo
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 11/66 | 11/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maxalt (N=66) | Placebo (N=66)
Chest tightness (Nervous system disorders) | 6 | 5 — Expected medication side effect
Heart palpitation (Nervous system disorders) | 4 | 6 — Expected medication side effect
Throat tightness (Nervous system disorders) | 7 | 4 — Expected medication side effect
Skin sensitivity (Nervous system disorders) | 6 | 3 — Expected medication side effect
Gastrointestinal (Nervous system disorders) | 8 | 3 — Expected medication side effect
Drowsiness (Nervous system disorders) | 9 | 1 — Expected medication side effect

LIMITATIONS AND CAVEATS:
Patients were not asked whether or not they thought the pill they took was maxalt or placebo. Thus, it is not possible to determine their actual level of expectation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No